CLINICAL TRIAL: NCT03568500
Title: A Multicentre, 8-week, Single-arm, Open-label, Pragmatic Trial to Explore Acceptance and Performance of Using a Digital Medicine System With Healthcare Professionals and Adult Subjects With Schizophrenia, Schizoaffective Disorder, or First Episode Psychosis on an Oral Atypical Antipsychotic (Aripiprazole, Olanzapine, Quetiapine, or Risperidone)
Brief Title: A Trial to Explore Acceptance and Performance of Using a Digital Medicine System With Healthcare Professionals and Adults With Schizophrenia, Schizoaffective Disorder, or First Episode Psychosis on an Oral Atypical Antipsychotic
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Development & Commercialization, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 031-201-00186
Record Dates: First submitted 2018-05-25; First posted 2018-06-26 (Actual); Results first posted 2020-07-16 (Actual); Last update posted 2020-07-16 (Actual); Status verified 2020-07

CONDITIONS: Schizophrenia; Schizoaffective Disorder; First Episode Psychosis
Keywords: Digital Medicine System
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — Aripiprazole; Olanzapine; Quetiapine Fumarate; Risperidone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Aripiprazole (Experimental): Participants received 1 oral tablet of CoEncapsulated (CoE) aripiprazole, wearing the DMS patch, and using the associated smartphone app for a total of 8 weeks.
  Interventions: Device: Digital Medicine System; Drug: Aripiprazole
- Olanzapine (Experimental): Participants received 1 oral tablet of CoE olanzapine, wearing the DMS patch, and using the associated smartphone app for a total of 8 weeks.
  Interventions: Device: Digital Medicine System; Drug: Olanzapine
- Quetiapine (Experimental): Participants received 1 oral tablet of CoE quetiapine, wearing the DMS patch, and using the associated smartphone app for a total of 8 weeks.
  Interventions: Device: Digital Medicine System; Drug: Quetiapine
- Risperidone (Experimental): Participants were to receive 1 oral tablet of CoE risperidone, wearing the DMS patch, and using the associated smartphone app for a total of 8 weeks. No participant took risperidone in this trial.
  Interventions: Device: Digital Medicine System; Drug: Risperidone

INTERVENTIONS:
Device: Digital Medicine System — DMS components: a CoE product consisting of an approved antipsychotic medicinal product co-encapsulated with Conformité Européenne (CE)-marked miniature ingestible event marker in tablet; a CE-marked compatible medical device (a Proteus Patch [Disposable Wearable Sensor Version 5]); proprietary medical software (a local and remote computing application).
Drug: Aripiprazole — Dosage determined by the healthcare professionals.
  Arms: Aripiprazole
Drug: Olanzapine — Dosage determined by the healthcare professionals.
  Arms: Olanzapine
Drug: Quetiapine — Dosage determined by the healthcare professionals.
  Arms: Quetiapine
Drug: Risperidone — Dosage determined by the healthcare professionals.
  Arms: Risperidone

SUMMARY:
Digital medicine systems (DMS) have been designed to assist individuals with the management of their daily health, wellness, and medication use. The DMS is being developed as a healthcare management tool to precisely measure medication adherence and to potentially enhance adherence.

DETAILED DESCRIPTION:
The advancements in the treatment of mental health patients with DMS will enable healthcare professionals to assess suboptimal adherence and make more informed treatment decisions. In addition to these improvements, it will also provide a platform for engagement between participants, healthcare professionals, and caregivers/support persons.

Participants who entered the trial were treated with one of the oral atypical antipsychotics defined in the trial (aripiprazole, olanzapine, quetiapine, or risperidone [though no participant took risperidone in this trial]). The treatment medication decision was determined by the healthcare professionals.

ELIGIBILITY:
Inclusion Criteria:

* Participant was prescribed aripiprazole, olanzapine, quetiapine, or risperidone.
* Participant possessed a smartphone, or a smartphone provided by the Sponsor, and was willing to download and interact with the DMS app.
* Skin on the anterior chest just above the lower edge of the rib cage was free of any dermatological problems (for example, open wounds, warts, rashes, atopic dermatitis).

Exclusion Criteria:

* Participant with a known allergy to adhesive tape or any pertinent components of the patch or CoE product.
* Prisoners could not be enrolled into this trial.
* Participant who was hospitalized due to mental or physical illness (inpatient) at the time of screening/baseline.
* Any participant who, through religious or lifestyle choices, would not take gelatin capsules.
* Female of childbearing potential who was breast-feeding and/or who had a positive pregnancy test result prior to receiving trial enrollment, or who planned to become pregnancy during the trial.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2018-05-21 (Actual); Primary Completion 2019-05-21 (Actual); Study Completion 2019-09-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (5):
- United Kingdom (5):
  - Clinical Trial Site, Chertsey
  - Clinical Trial Site, London
  - Clinical Trial Site, Newcastle upon Tyne
  - Clinical Trial Site, Oxford
  - Clinical Trial Site, Southampton

IPD SHARING:
Plan to Share IPD: Yes
Anonymized Individual participant data (IPD) that underlie the results of this study will be shared with researchers to achieve aims pre-specified in a methodologically sound research proposal. Small studies with less than 25 participants are excluded from data sharing.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data will be available after marketing approval in global markets, or beginning 1-3 years following article publication. There is no end date to the availability of the data.
Access Criteria: Otsuka will share data on an Otsuka-owned remotely accessible data sharing platform with Python and R analytical software. Research requests should be directed to clinicaltransparency@Otsuka-us.com.
URL: https://clinical-trials.otsuka.com

REFERENCES:
- [Derived] Jan M, Coppin-Renz A, West R, Gallo CL, Cochran JM, Heumen EV, Fahmy M, Reuteman-Fowler JC. Safety Evaluation in Iterative Development of Wearable Patches for Aripiprazole Tablets With Sensor: Pooled Analysis of Clinical Trials. JMIR Form Res. 2023 Dec 12;7:e44768. doi: 10.2196/44768. PMID 38085556
- [Derived] Fowler JC, Cope N, Knights J, Phiri P, Makin A, Peters-Strickland T, Rathod S. Hummingbird Study: a study protocol for a multicentre exploratory trial to assess the acceptance and performance of a digital medicine system in adults with schizophrenia, schizoaffective disorder or first-episode psychosis. BMJ Open. 2019 Jun 27;9(6):e025952. doi: 10.1136/bmjopen-2018-025952. PMID 31253613

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial enrolled participants with a confirmed clinical diagnosis of schizophrenia, schizoaffective disorder, or first episode psychosis.
Pre-assignment Details: Participants in this trial received at least 1 CoEncapsulated miniature ingestible event marker in a tablet and a medicinal product originator tablet of either aripiprazole, olanzapine, or quetiapine (participants were allowed to take risperidone, though no participant took risperidone in this trial) as prescribed by their healthcare professional.
Groups:
- Aripiprazole: Participants were treated with at least 1 CoEncapsulated (CoE) oral aripiprazole tablet, wearing the digital medicine system (DMS) patch, and using the associated smartphone app for a total of 8 weeks.
- Olanzapine: Participants were treated with at least 1 CoE oral olanzapine tablet, wearing the DMS patch, and using the associated smartphone app for a total of 8 weeks.
- Quetiapine: Participants were treated with at least 1 CoE oral quetiapine tablet, wearing the DMS patch, and using the associated smartphone app for a total of 8 weeks.
Period: Overall Study
Arm/Group | Aripiprazole | Olanzapine | Quetiapine
Started | 18 | 20 | 6
Received At Least 1 Dose of Study Drug (Safety Population: All participants who entered the trial and used the DMS.) | 18 | 19 | 6
Completed | 8 | 14 | 2
Not Completed | 10 | 6 | 4
Not completed — Lost to Follow-up | 1 | 1 | 2
Not completed — Adverse Event | 1 | 1 | 2
Not completed — Physician Decision | 1 | 0 | 0
Not completed — Withdrawal by Subject | 4 | 2 | 0
Not completed — Technical Problems | 2 | 1 | 0
Not completed — Participant Noncompliance | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Enrolled Population: All participants who signed an informed consent form and entered the trial (and only participants who met all of the inclusion criteria and none of the exclusion criteria).
Groups:
- Total: Total of all reporting groups
Arm/Group | Aripiprazole | Olanzapine | Quetiapine | Total
Number analyzed (Participants) | 18 | 20 | 6 | 44
Age, Continuous [Mean (Standard Deviation); unit: Years] | 31.6 (9.6) | 38.0 (11.4) | 30.8 (8.8) | 34.4 (10.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 4 | 3 | 15
  Male | 10 | 16 | 3 | 29
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 17 | 18 | 5 | 40
  Unknown or Not Reported | 1 | 2 | 1 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 4 | 4 | 0 | 8
  White | 14 | 15 | 6 | 35
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 0 | 1
Disease Diagnosis [Count of Participants; unit: Participants]
  Schizophrenia | 5 | 13 | 0 | 18
  Schizoaffective Disorder | 4 | 4 | 2 | 10
  First Episode Psychosis | 9 | 3 | 4 | 16

OUTCOME MEASURES:

1. Primary Outcome: Percentage Of Days With Good Patch Coverage
Description: The DMS includes a drug-device combination of a CoE product, a wearable sensor patch, and application software (smartphone) to record activity and rest and mark events through the act of ingestion. The CoE product consists of an approved antipsychotic medication enclosed with an Ingestible Sensor Pill (miniature ingestible event marker in tablet [MIT]). The sensor patch detects and records each MIT ingestion, as well as other physiologic and behavioral data. Good patch coverage for a specific day was defined as having either at least 80% patch data available (80% of the day the patch was worn and data was collected as noted via the accelerometer channel) or the MIT was detected within the 24-hour period, for each day while the participant was in the trial. The percentage of days was calculated as the number of days with good patch coverage divided by the total number of trial days for each participant. Descriptive statistics were performed for this outcome measure.
Time Frame: Up to 8 weeks
Population: Intent-to-treat (ITT) Population: All participants who entered the trial and used the DMS.
Measure: Mean (Standard Deviation); unit: percentage of days
Groups:
- Schizophrenia: Participants had a confirmed clinical diagnosis of schizophrenia (defined by International Classification of Disease-10 codes F20 and F25). There was no limit on the duration of illness. Participants were treated with at least 1 CoE oral atypical antipsychotic tablet (aripiprazole, olanzapine, or quetiapine), wearing the DMS patch, and using the associated smartphone app for a total of 8 weeks. The treatment medication decision was determined by the healthcare professional.
- Schizoaffective Disorder: Participants had a confirmed clinical diagnosis of schizoaffective disorder (defined by International Classification of Disease-10 codes F20 and F25). There was no limit on the duration of illness. Participants were treated with at least 1 CoE oral atypical antipsychotic tablet (aripiprazole, olanzapine, or quetiapine), wearing the DMS patch, and using the associated smartphone app for a total of 8 weeks. The treatment medication decision was determined by the healthcare professional.
- First Episode Psychosis: Participants had a confirmed clinical diagnosis of first episode psychosis using case note review. The duration of illness was defined as less than 3 years since presentation to the mental health team or first antipsychotic prescription. Participants were treated with at least 1 CoE oral atypical antipsychotic tablet (aripiprazole, olanzapine, or quetiapine), wearing the DMS patch, and using the associated smartphone app for a total of 8 weeks. The treatment medication decision was determined by the healthcare professional.
- Total: Participants were treated with at least 1 CoE oral atypical antipsychotic tablet (aripiprazole, olanzapine, or quetiapine), wearing the DMS patch, and using the associated smartphone app for a total of 8 weeks. The treatment medication decision was determined by the healthcare professional.
Arm/Group | Schizophrenia | Schizoaffective Disorder | First Episode Psychosis | Total
Number analyzed (Participants) | 18 | 9 | 16 | 43
percentage of days | 64.34 (20.24) | 62.99 (37.68) | 62.51 (27.53) | 63.37 (26.60)

2. Secondary Outcome: Participant Adherence
Description: The DMS includes a drug-device combination of a CoE product, a wearable sensor patch, and application software (smartphone) to record activity and rest and mark events through the act of ingestion. The CoE product consists of an approved antipsychotic medication enclosed with an Ingestible Sensor Pill (MIT). The sensor patch detects and records each MIT ingestion, as well as other physiologic and behavioral data. Participant adherence was measured as the detected MITs over the expected MITs ingested during the trial days with good patch coverage. The more the participant successfully engaged in a number of processes across the 8-week trial, the greater the measured adherence. Descriptive statistics were performed for this outcome measure.
Time Frame: Up to 8 weeks
Population: Intent-to-treat (ITT) Population: All participants who entered the trial, used the DMS, and had data available at the specified timepoint.
Measure: Mean (Standard Deviation); unit: percentage of MITs
Groups:
- Schizophrenia: Participants had a confirmed clinical diagnosis of schizophrenia (defined by International Classification of Disease-10 codes F20 and F25). There was no limit on the duration of illness. Participants were treated with at least 1 CoE oral atypical antipsychotic tablet (aripiprazole, olanzapine, or quetiapine), wearing the DMS patch, and using the associated smartphone app for a total of 8 weeks. The treatment medication decision was determined by the HCP.
- Schizoaffective Disorder: Participants had a confirmed clinical diagnosis of schizoaffective disorder (defined by International Classification of Disease-10 codes F20 and F25). There was no limit on the duration of illness. Participants were treated with at least 1 CoE oral atypical antipsychotic tablet (aripiprazole, olanzapine, or quetiapine), wearing the DMS patch, and using the associated smartphone app for a total of 8 weeks. The treatment medication decision was determined by the HCP.
- First Episode Psychosis: Participants had a confirmed clinical diagnosis of first episode psychosis using case note review. The duration of illness was defined as less than 3 years since presentation to the mental health team or first antipsychotic prescription. Participants were treated with at least 1 CoE oral atypical antipsychotic tablet (aripiprazole, olanzapine, or quetiapine), wearing the DMS patch, and using the associated smartphone app for a total of 8 weeks. The treatment medication decision was determined by the HCP.
Arm/Group | Schizophrenia | Schizoaffective Disorder | First Episode Psychosis | Total
Number analyzed (Participants) | 18 | 8 | 16 | 42
percentage of MITs | 88.94 (8.06) | 72.29 (25.65) | 91.04 (7.37) | 86.57 (14.47)

ADVERSE EVENTS:
Time Frame: Baseline to Week 24 (+ 7 days)
Arm/Group | Aripiprazole | Olanzapine | Quetiapine | Total
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/19 | 0/6 | 0/43
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/19 | 0/6 | 0/43
Other Adverse Events (participants affected / at risk) | 4/18 | 2/19 | 3/6 | 9/43
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Aripiprazole (N=18) | Olanzapine (N=19) | Quetiapine (N=6) | Total (N=43)
Medical device site irritation (General disorders) | 4 (5) | 2 (2) | 3 (4) | 9 (11)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right to review results publications prior to public release and can delay such publications for a period greater than 60 days but no more than 120 days from the date that the publication is submitted to the Sponsor for review. Sponsor can require changes to the publication to protect Sponsor's intellectual property rights and/or confidential information and reserves the right to limit publication timing and scope of data published based on the number of study locations.

DOCUMENTS (3):
  • Study Protocol: Version 1.0 (2017-12-01): https://cdn.clinicaltrials.gov/large-docs/00/NCT03568500/Prot_000.pdf
  • Study Protocol: Version 2.0 (2019-01-04): https://cdn.clinicaltrials.gov/large-docs/00/NCT03568500/Prot_001.pdf
  • Statistical Analysis Plan (2019-06-30): https://cdn.clinicaltrials.gov/large-docs/00/NCT03568500/SAP_002.pdf